CLINICAL TRIAL: NCT05262140
Title: In Vivo Quantification of Cervical Collar Efficacy
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 071.TRA.2021.D
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Spine Injury
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective interventional trial with healthy volunteers at Methodist Dallas Medical Center. We anticipate data collection to be completed by December 2023. All study participants will be consented regardless of their role as healthy C-spine volunteer or provider volunteer (Appendix C). No compensation will be provided. Provider volunteers will be classified as:

* Attending
* Resident
* Physician assistant, nurse practitioner, or nurse
* EMS/Paramedic
* Other, as determined by job functions in pre-assessment

DETAILED DESCRIPTION:
This is a prospective interventional trial with healthy volunteers at Methodist Dallas Medical Center. We anticipate data collection to be completed by December 2023. All study participants will be consented regardless of their role as healthy C-spine volunteer or provider volunteer (Appendix C). No compensation will be provided. Provider volunteers will be classified as:

* Attending
* Resident
* Physician assistant, nurse practitioner, or nurse
* EMS/Paramedic
* Other, as determined by job functions in pre-assessment Prior to placing C-collars, provider volunteers who will be placing C-collars will answer a questionnaire about their medical experience, their current position, their confidence in effective C-collar placement, and if they had formal C-collar training (Appendix D).

Healthy C-spine volunteers will lie supine. Cameras will be placed directly superior, anterior, and lateral to the volunteer's head. C-spine volunteers will be asked to actively move their head to the maximal flexion, extension, bilateral rotation, and bilateral side bending to assess baseline ROM.

Provider volunteers will individually place a C-collar on the C-spine volunteer's neck. They will have a range of sizes to choose from or adjustable units as applicable. The provider volunteer will be able to independently select and adjust a collar to best fit the C-spine volunteer.

The C-spine volunteer will then actively move their head to the maximal flexion, extension, bilateral rotation, and bilateral side bending with the C-collar on. ROM will be analyzed from video taken. This process will be repeated for each C-spine volunteer and each provider volunteer (Minimum 3 volunteers per 1 provider volunteer).

The angle of ROM in flexion, extension, rotation, and side bending without and with C-collar placement in each video will be measured using image analysis software. The decrease in ROM while wearing the C-collar for each encounter will be calculated. Scoring of C-collar placement will be done by an investigator while the provider volunteer is placing the C-collar. Providers will then receive additional information and resources specific to C-collar make/model placement and asked to complete a short survey (Appendix E) related to the content provided.

Provider volunteers will then have training on correct sizing and placing of C-collars and be reassessed in the same manor described above. Percent change will then be calculated for each volunteer provider.

This is a prospective interventional trial with healthy volunteers at Methodist Dallas Medical Center. We anticipate data collection to be completed by December 2023. All study participants will be consented regardless of their role as healthy C-spine volunteer or provider volunteer (Appendix C). No compensation will be provided. Provider volunteers will be classified as:

* Attending
* Resident
* Physician assistant, nurse practitioner, or nurse
* EMS/Paramedic
* Other, as determined by job functions in pre-assessment Prior to placing C-collars, provider volunteers who will be placing C-collars will answer a questionnaire about their medical experience, their current position, their confidence in effective C-collar placement, and if they had formal C-collar training (Appendix D).

Healthy C-spine volunteers will lie supine. Cameras will be placed directly superior, anterior, and lateral to the volunteer's head. C-spine volunteers will be asked to actively move their head to the maximal flexion, extension, bilateral rotation, and bilateral side bending to assess baseline ROM.

Provider volunteers will individually place a C-collar on the C-spine volunteer's neck. They will have a range of sizes to choose from or adjustable units as applicable. The provider volunteer will be able to independently select and adjust a collar to best fit the C-spine volunteer.

The C-spine volunteer will then actively move their head to the maximal flexion, extension, bilateral rotation, and bilateral side bending with the C-collar on. ROM will be analyzed from video taken. This process will be repeated for each C-spine volunteer and each provider volunteer (Minimum 3 volunteers per 1 provider volunteer).

The angle of ROM in flexion, extension, rotation, and side bending without and with C-collar placement in each video will be measured using image analysis software. The decrease in ROM while wearing the C-collar for each encounter will be calculated. Scoring of C-collar placement will be done by an investigator while the provider volunteer is placing the C-collar. Providers will then receive additional information and resources specific to C-collar make/model placement and asked to complete a short survey (Appendix E) related to the content provided.

Provider volunteers will then have training on correct sizing and placing of C-collars and be reassessed in the same manor described above. Percent change will then be calculated for each volunteer provider.

ELIGIBILITY:
Inclusion Criteria:

C-spine Volunteers:

* Methodist Dallas Medical Center (MDMC) staff
* 18+ years old
* Full ROM of C-spine

Provider Volunteers:

* Medical provider with permissions at MDMC
* C-collar placement in regular job duties

Exclusion Criteria:

* C-spine Volunteers:

  * <18 years old
  * C-spine trauma
  * Previous neck or C-spine surgeries
  * Abnormal limitations to C-spine ROM
  * Pregnant/nursing
  * Claustrophobia
  * Pulmonary dysfunction

Provider Volunteers:

• No previous experience placing C-collars

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective interventional trial with healthy volunteers at Methodist Dallas Medical Center. We anticipate data collection to be completed by December 2023. All study participants will be consented regardless of their role as healthy C-spine volunteer or provider volunteer (Appendix C). No compensation will be provided. Provider volunteers will be classified as:
  * Attending
  * Resident
  * Physician assistant, nurse practitioner, or nurse
  * EMS/Paramedic
  * Other, as determined by job functions in pre-assessment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2025-01-19 (Estimated); Study Completion 2025-01-19 (Estimated)

PRIMARY OUTCOMES:
placement of a c-collar | Dec 2021 - Dec 2022
  Each volunteer provider will be scored on their placement of a c-collar before and after review of educational materials based on the fit criteria provided by the C-collar manufacturer.
Measurements will be taken from videos captured | Dec 2021 - Dec 2022
  Measurements will be taken from videos captured during the study. Image analysis software will be used to measure the angles of motion for each
Percent change in the angle of ROM | Dec 2021 - Dec 2022
  Percent change in the angle of ROM in flexion, extension, rotation, and side bending with and without C-collar placement.

CONTACTS AND LOCATIONS:
Overall Officials: Conner McDaniel, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States